CLINICAL TRIAL: NCT04144634
Title: Pilot Study of an Exercise Programme to Maintain Knee Extension Muscle Strength for Older Patients During Hospitalisation
Brief Title: Feasibility of Additional Physiotherapy for Patients Aged 75 and Older
Acronym: Stand-UP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to COVID-19
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other); University of Dublin, Trinity College (Other); The Dunhill Medical Trust (Other); Addenbrooke's Charitable Trust (Unknown)
Responsible Party: Principal Investigator, Peter Hartley, Physiotherapist, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A095191; 252802 (Other: IRAS)
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Exercise; Hospitalisation; Older Adults
MeSH Terms: conditions — Motor Activity | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention/Strengthening (Experimental)
  Interventions: Other: Strengthening exercises
- Control/Stretching (Sham Comparator)
  Interventions: Other: Stretching exercises

INTERVENTIONS:
Other: Strengthening exercises — The intervention group will receive 2 supervised exercise sessions a day. The exercise consists of progressive resistance training based around the movement of standing up/sitting down.
  Arms: Intervention/Strengthening
Other: Stretching exercises — The intervention group will receive 2 supervised exercise sessions a day. The exercise consists of gentle stretching of upper limbs and lower limbs.
  Arms: Control/Stretching

SUMMARY:
On average, people become physically weaker during even a short stay in hospital. This study is a feasibility/pilot study to see if additional physiotherapy exercises undertaken in hospital is feasible and acceptable to patients.

The study will compare two different types of physiotherapy exercise. Both exercise programmes involve twice-daily physiotherapy provided by one of the hospital's physiotherapy assistants, but only one of the two exercise programmes expected to provide benefit. This is on top of the care that people would normally receive, and will last for the first 7 days of their hospital admission (or until they are discharged if this is earlier).

Patients will be asked to consent to the study during the first 36 hours of their hospital admission. If patients provide consent, they will undergo a baseline assessment of their functional ability (including testing of their muscle strength) before being randomly assigned to one of the two exercise programmes. The study aims to recruit 15 patients to each group (30 in total).

Once randomised patients will be seen twice a day by a physiotherapy assistant who will supervise the exercise programme.

On the day that participants are discharged (or day 7 of their admission if earlier) the assessor will repeat measures of the participants functional ability. Following these measures participants will be invited to be interviewed to discuss their experience of taking part in the study.

Approximately one month after discharge, a researcher will visit the participant to repeat measures of their functional ability at their home.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to CUH, who are aged 75 or older, able to give informed consent and expected to be hospitalised more than 24 hours.

Exclusion Criteria:

* Admitted more than 36 hours prior to recruitment; unable to provide informed consent (e.g. due to dementia, delirium, cognitive impairment); receiving end of life care or oncological treatment for diagnosed cancer; inability to cooperate in muscle strength testing (e.g. unable to sit in chair, or presence of skin integrity problems contraindicating the use of a hand-held dynamometer); transferred to or from the intensive care unit; bed-bound or requiring a hoist to transfer from bed to chair 2 weeks prior to hospitalisation; or if the Consultant in charge of the patient has any other clinical concerns regarding participation in a strengthening exercise programme.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Topic-guided interview of participants at discharge from hospital | At day 7 of hospitalisation (or at discharge if earlier)

SECONDARY OUTCOMES:
Topic-guided semi-structured interview of the group of physiotherapy assistants who delivered the intervention | At day 7 of hospitalisation (or at discharge if earlier)
Hand held dynamometry (Knee extension + grip strength) | At day 7 of hospitalisation (or at discharge if earlier), follow up 6 weeks after discharge
de Morton Mobility Index | At day 7 of hospitalisation (or at discharge if earlier), follow up 6 weeks after discharge
  Scale from 0-100, 100 representing highest functional ability
Barthel Index | 6 weeks after discharge
  Scale from 0-100, 100 representing highest functional ability
Falls Efficacy Scale International | 6 weeks after discharge
  Scale from 16-64, 16 representing highest perceived self efficacy of avoiding falling
Confidence measured on a visual analogue scale | 6 weeks after discharge
  Scale from 0-100, 100 representing highest level of confidence.
Mini-Addenbrookes Cognitive Examination | 6 weeks after discharge
  Scale from 0-30, 30 representing highest cognitive ability.
Survey of Health, Ageing and Retirement in Europe (SHARE) Frailty Instrument | 6 weeks after discharge
  A continuous scale, with a higher number representing a higher degree of frailty
Physical activity in hospital | 6 weeks after discharge
  Measured with accelerometers

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No